CLINICAL TRIAL: NCT02299674
Title: Investigation of Medial Lateral Displacement of Center of Pressure and Center of Mass During Double Support in Men With Unilateral Transfemoral Amputations.
Brief Title: Study of Medial-Lateral Center of Pressure Displacement in Unilateral Transfemoral Amputees
Status: Completed | Type: Observational
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Dana Craig, Health System Specialist, Southern California Institute for Research and Education
Other Study IDs: 1316
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Unilateral Transfemoral Amputation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Persons with unilateral transfemoral amputation
  Interventions: Other: Level overground ambulation

INTERVENTIONS:
Other: Level overground ambulation

SUMMARY:
The purpose of this study is to examine the path and velocity of the center of mass (CoM) and center of pressure (CoP) during double support of persons walking with a unilateral above-the-knee prosthesis and determine the effects of prosthetic foot stiffness and effective length on CoM and CoP.Persons with a lower limb amputation walk with compensatory movements that affect the smooth trajectory of the center of mass (CoM) during weight transfer. The lack of control in the foot/ankle complex reduces fine motor movements, influencing the progression of the CoM and transfer of ground reaction forces represented by the center of pressure (CoP). Without control of the ankle joint, prosthetic users "fall" off of their trailing prosthetic limb during weight transfer, resulting in much more abrupt CoM and CoP transfers from trailing to leading limb. These abrupt movements during transfer not only increase stress on the sound limb, but also decrease the subject's energy efficiency during ambulation. The current study will further examine the CoP path and velocity in relation to the CoM path and velocity during double support of men with a transfemoral prosthesis, as well as explore how prosthetic foot ankle stiffness and effective length affects the CoP path and velocity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a transfermoral amputation and use an above-the-knee prosthesis with an articulating knee joint on a daily basis.
* Participants must be male.
* Age greater than or equal to 18 years, but less than 65 years.
* Participants must have no known pathology or comorbidites that would affect their ambulatory ability
* Ability to tolerate walking for a minimum of 100 yards over the course of a two and a half hour time period.
* Ability to walk one block without needing to rest.

Exclusion Criteria:

* Use of ambulatory aids such as canes or crutches.
* Any medical or psychosocial condition that, in the opinion of the investigator, could jeopardize the subject's participation, and compliance with the study criteria.
* Bilateral amputations.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with unilateral transfemoral amputation who are ambulatory with a prosthesis and no assistive device.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Center of Pressure Velocity | Double Support Phase of Gait Cycle (2.5 hour)
  The Center of Pressure velocity in the X and Y direction [cm/sec] will be collected using a motion capture system and forceplates during a single session. This data will be collected during a single 2.5 hour data collection session. The time frame is specifically the Double Support phase of the gait cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- V.A. Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Au, S. K., Weber, J., & Herr, H. (2009). Powered Ankle-Foot Prosthesis Improves Walking Metabolic Economy. IEEE Transactions on Robotics, 25(1), 51-66.
- [Background] Donelan JM, Kram R, Kuo AD. Simultaneous positive and negative external mechanical work in human walking. J Biomech. 2002 Jan;35(1):117-24. doi: 10.1016/s0021-9290(01)00169-5. PMID 11747890
- [Background] Herr HM, Grabowski AM. Bionic ankle-foot prosthesis normalizes walking gait for persons with leg amputation. Proc Biol Sci. 2012 Feb 7;279(1728):457-64. doi: 10.1098/rspb.2011.1194. Epub 2011 Jul 13. PMID 21752817
- [Background] Hof AL, van Bockel RM, Schoppen T, Postema K. Control of lateral balance in walking. Experimental findings in normal subjects and above-knee amputees. Gait Posture. 2007 Feb;25(2):250-8. doi: 10.1016/j.gaitpost.2006.04.013. Epub 2006 Jun 5. PMID 16740390
- [Background] Kadaba MP, Ramakrishnan HK, Wootten ME. Measurement of lower extremity kinematics during level walking. J Orthop Res. 1990 May;8(3):383-92. doi: 10.1002/jor.1100080310. PMID 2324857
- [Background] Nolan KJ, Yarossi M. Weight transfer analysis in adults with hemiplegia using ankle foot orthosis. Prosthet Orthot Int. 2011 Mar;35(1):45-53. doi: 10.1177/0309364610393061. PMID 21515889
- [Background] Orendurff MS, Segal AD, Klute GK, Berge JS, Rohr ES, Kadel NJ. The effect of walking speed on center of mass displacement. J Rehabil Res Dev. 2004 Nov-Dec;41(6A):829-34. doi: 10.1682/jrrd.2003.10.0150. PMID 15685471
- [Background] Schmid M, Beltrami G, Zambarbieri D, Verni G. Centre of pressure displacements in trans-femoral amputees during gait. Gait Posture. 2005 Apr;21(3):255-62. doi: 10.1016/j.gaitpost.2004.01.016. PMID 15760740
- [Background] Turnbull GI, Charteris J, Wall JC. Deficiencies in standing weight shifts by ambulant hemiplegic subjects. Arch Phys Med Rehabil. 1996 Apr;77(4):356-62. doi: 10.1016/s0003-9993(96)90084-2. PMID 8607759